CLINICAL TRIAL: NCT06510257
Title: Safety and Efficacy of Reconyl for Cough With/Without Sore Throat: A Preliminary Study
Brief Title: Safety and Efficacy Reconyl for Cough With/Without Sore Throat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRSU.P.Dexa/06/20/10.03A
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cough
Keywords: Cough with sore throat; Cough without sore throat; Reconyl
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): 1 tablet of Reconyl, 3 times daily
  Interventions: Drug: Reconyl
- Control Group (Placebo Comparator): 1 tablet of placebo Reconyl, 3 times daily
  Interventions: Drug: Placebo tablet of Reconyl

INTERVENTIONS:
Drug: Reconyl — 1 tablet of Reconyl, 3 times daily
  Other Names: HerbaKOF
  Arms: Treatment Group
Drug: Placebo tablet of Reconyl — 1 tablet of placebo Reconyl, 3 times daily
  Arms: Control Group

SUMMARY:
This study is a prospective, randomized, double-blind and placebo-controlled study to find out if reconyl may relieve the acute cough with/without sore throat.

DETAILED DESCRIPTION:
Reconyl is a mixed extract from 4 Indonesian herbs, Vitex trifolia (Legundi), Zingiber officinale var. Amarum (Jahe Gajah), Abrus precatorius (Saga), and Phaleria macrocarpa (Mahkota Dewa), which have been known traditionally to relieve cough, respiratory congestion, and sore throat.

There will be two parallel groups of 30 subjects per group (a total of 60 subjects) planned to be enrolled in this study.

The investigational product: tablets @ 225 mg of Reconyl. Dose administration: One tablet of Reconyl or Placebo, given 3 times daily, for 3 days.

Eligible subjects will be instructed to perform a daily self-assessment on the cough symptoms over the 3 days of treatment, in the Subject Diary. Subject shall return to the study clinic 3 days ± 24 hours after the first dose, for completion of the subject's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women aged 18 to 60 years with cough with/without sore throat with a maximum onset of 3 days.
2. Signing the informed consent.

Exclusion Criteria:

1. Body temperature of > 37.3˚C and/or refuse to follow health protocol for COVID-19
2. Known hypersensitivity to herbal drugs
3. Pregnant or lactating women
4. Have received any anti-inflammatory or cough-alleviating drugs within the past 24 hours
5. Presence of vomiting or diarrhea within the past 24 hours and still ongoing at the start of study
6. Severe illness, e.g. severe hypertension, any other chronic infections or diseases that may induce cough, such as: pulmonary tuberculosis, gastrointestinal reflux diseases (GERD)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Cough score | Day 0, Day 1, Day 2, Day 3
  Scoring will be performed and recorded daily in the Subject Diary at time 0, every night time and before the morning dose.
  At the End of Study (last visit) will be assessed by the subject and recorded by the Investigator.
  Cough score:
  • Day time: 0 = No cough; 1= Transient cough occasionally during the daytime; 2 = Frequent cough mildly affecting daily life; 3 = Frequent cough severely affecting daily life.
  • Night time: 0 = No cough; 1= Transient cough before sleep or occasional cough during the night; 2 = Cough mildly affecting night sleep; 3 = Cough severely affecting night sleep.
Visual Analogue Scale (VAS) | Day 0, Day 1, Day 2, Day 3
  Visual Analogue Scale (VAS) for sore throat (0 - 100), with 0 indicates asymptomatic and 100 refers to the most serious or severe symptom.
  VAS will be assessed and recorded daily in Subject Diary at time 0, every night time and before the morning dose.
  At the End of Study (last visit) will be assessed by the subject and recorded by the Investigator.
Adverse events | Day 0, Day 1, Day 2, Day 3
  Any adverse events (AE) and serious adverse events (SAE) will be observed throughout the study conduct.

CONTACTS AND LOCATIONS:
Overall Officials: Dewi S Rosdiana, Dr,MD,MKes, Principal Investigator — Department Pharmacology & Therapeutics Faculty of Medicine Universitas Indonesia
Locations (2):
- Indonesia (2):
  - Imeri Fkui, Jakarta Pusat, DKI Jakarta
  - Klinik Satelit Makara UI Depok, Depok, West Java